CLINICAL TRIAL: NCT03596944
Title: Primary Prevention With Statin and Incidence of Recurrent Myocardial Infarction and Cardiogenic Shock in Post-Acute Coronary Syndrome Patients
Brief Title: Primary Prevention With Statin and Incidence of Recurrent MI and Cardiogenic Shock in Post-ACS Patients
Status: Completed | Type: Observational
Sponsor: Tarumanagara University (Other)
Collaborators: Cengkareng General Hospital (Other)
Responsible Party: Principal Investigator, Angela Felicia Sunjaya, Principal Investigator, Tarumanagara University
Other Study IDs: APS005
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome; Recurrent Myocardial Infarction; Cardiogenic Shock
Keywords: acute coronary syndrome; statin; mortality; GRACE score; TIMI score
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Shock, Cardiogenic | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin: History of statin use for primary prevention
  Interventions: Drug: Statin
- Non-Statin: No documented history of statin use prior to Acute Coronary Syndrome

INTERVENTIONS:
Drug: Statin — Prescribed with statins for primary prevention
  Groups: Statin

SUMMARY:
This study aims to evaluate the effect of statin for primary prevention, towards lowering the incidence of recurrent myocardial infarction, cardiogenic shock and mortality in ACS patients.

DETAILED DESCRIPTION:
Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under ICD-10 coding of I24.9 were included in this study. The inclusion criteria are patients with primary diagnosis of I24.9 and with a complete record of prior medical and treatment history, electrocardiographic findings, cardiac marker results and outcomes. Participants were grouped into 2 groups - statin and non-statin based on prior history of statin use prior to ACS. Diagnosis of ACS was made based on clinical, electrocardiographic and cardiac marker findings found in the medical record.

Data such as age, sex, ethnic, education, prior medical and treatment history, electrocardiographic and cardiac enzyme results as well as outcomes were collected from the patients' medical records. Outcomes of interest were defined as either recurrent myocardial infarction, cardiogenic shock, mortality or combinations of them as diagnosed in the medical records. GRACE and TIMI Scores are calculated to predict in hospital and future mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Coronary Syndrome
* Presence of detail on statin prescription history

Exclusion Criteria:

* Unavailability of electrocardiographic findings, cardiac marker results, GRACE and TIMI score parameters
* Incomplete records of prior medical and treatment history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under International Classification of Diseases (ICD)10 coding of I24.9
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Recurrent Myocardial Infarction | Through study completion, an average of 1 year
  Clinical Diagnosis of Recurrent Myocardial Infarction reported in medical records
Cardiogenic Shock | Through study completion, an average of 1 year
  Clinical Diagnosis of Cardiogenic Shock reported in medical records
Mortality | Through study completion, an average of 1 year
  Patient death reported in medical records

OTHER OUTCOMES:
GRACE Score | Through study completion, an average of 1 year
  GRACE (Global Registry of Acute Coronary Events) mortality risk score
TIMI Score | Through study completion, an average of 1 year
  Thrombolysis In Myocardial Infarction (TIMI) mortality risk score

CONTACTS AND LOCATIONS:
Overall Officials: Angela F Sunjaya, Study Chair — Tarumanagara University; Anthony P Sunjaya, Principal Investigator — Tarumanagara University; Andria Priyana, MD, FIHA, Principal Investigator — Department of Cardiology, Faculty of Medicine, Tarumanagara University
Locations (1):
- Cengkareng General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided